CLINICAL TRIAL: NCT04536376
Title: First Responder Resiliency Program for Health Care Professionals During a Pandemic
Brief Title: First Responder Resiliency Program During COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: PNMedical (Industry)
Responsible Party: Principal Investigator, Ivana T Croghan, PhD, Professor of Medicine, College of Medicine, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-005017
Record Dates: First submitted 2020-08-26; First posted 2020-09-02 (Actual); Results first posted 2024-05-13 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2023-12

CONDITIONS: Resilience; Stress; Sleep

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Resilience Program (Experimental): a 4 week program focused on improving resilience
  Interventions: Behavioral: Resilience Program

INTERVENTIONS:
Behavioral: Resilience Program — Subjects receive program devices, and will be asked to wear during rest and sleep on a nightly basis along with active use during daytime. Notifications are sent daily, individualized approach developed and sent to participants to participate on.

SUMMARY:
Evaluating a wellness program developed to provide effective sustainable solutions for medical professionals providing care to COVID-19 pandemic patients.

DETAILED DESCRIPTION:
Providing mindfulness training at specific time points during study participation with an emphasis on integrating physical and mental health management. The phase-based program delivers individualized, data-driven and quantifiable solutions that directly address pain points impacting healthcare professionals and organizations.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older at the time of consent
2. Frontline healthcare professional
3. Have access to an Apple or Android device
4. Not pregnant by subject self-report at time of consent
5. Have the ability to provide informed consent
6. Have no contraindicating comorbid health condition as determined by the clinical investigators

Exclusion Criteria:

1. Currently (within the past 3 weeks) been practicing mindfulness training on a weekly/regular basis
2. Currently (within the past 3 weeks) been undergoing an additional program (e.g. CAM) to improve quality of life or sleep
3. Currently (within 3 weeks) been enrolled in another clinical or research program (e.g. CAM) which intervenes on the patients' QOL, stress or sleep
4. An unstable medical or mental health condition as determined by the physician investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-09-02 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivana T Croghan, PhD, Principal Investigator — Mayo Clinic; Brent Bauer, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Croghan IT, Hurt RT, Fokken SC, Fischer KM, Lindeen SA, Schroeder DR, Ganesh R, Ghosh K, Bausek N, Bauer BA. Stress Resilience Program for Health Care Professionals During a Pandemic: A Pilot Program. Workplace Health Saf. 2023 Apr;71(4):173-180. doi: 10.1177/21650799221093775. Epub 2022 Jul 5. PMID 35787711
- See also: Citation link — https://pubmed.ncbi.nlm.nih.gov/35787711/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Resilience Program
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Resilience Program
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.7 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Perceived Stress Scale
Description: Perceived Stress Scale (PSS) is a 10-item Likert scale scoring system that measures global life stress by assessing the degree to which experiences are appraised as uncontrollable or unpredictable. Scores can range from 0 to 40, with higher scores indicating greater perceived stress. The outcome was analyzed as change from baseline
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Resilience Program
Number analyzed (Participants) | 10
units on a scale | -3.2 (3.9)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Resilience Program
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/76/NCT04536376/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/76/NCT04536376/SAP_001.pdf